CLINICAL TRIAL: NCT04801888
Title: A Study to Evaluate the Safety and Immunogenicity of Concomitant Administration of the SARS-CoV-2 Inactivated Vaccine (Vero Cell) With Quadrivalent Influenza Vaccine in Adults Aged From 18 to 59 Years
Brief Title: Study on Combined Vaccination With SARS-CoV-2 Inactivated Vaccine and Quadrivalent Influenza Vaccine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sinovac Research and Development Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Sinovac Biotech Co., Ltd (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PRO-QINF-4001
Record Dates: First submitted 2021-03-15; First posted 2021-03-17 (Actual); Last update posted 2021-07-26 (Actual); Status verified 2021-03

CONDITIONS: COVID-19; Influenza
MeSH Terms: conditions — COVID-19; Influenza, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Combined immunization group (Experimental): The combined immunization group is randomly divided into two subgroups, 120 subjects in each group. The combined immunization subgroup Ⅰ receive SARS-CoV-2 inactivated vaccine (Vero cell)&Quadrivalent Influenza Vaccine on day0 and SARS-CoV-2 inactivated vaccine (Vero cell) (second dose) on day 28.The combined immunization subgroup Ⅱ receive SARS-CoV-2 inactivated vaccine (Vero cell) on day 0 and SARS-CoV-2 inactivated vaccine (Vero cell) (second dose) & Quadrivalent Influenza Vaccine on day 28.
  Interventions: Biological: Two doses of inactivated SARS-CoV-2 vaccine at the schedule of day 0,28 and one dose Quadrivalent Influenza Vaccine on day 0 or day 28.
- Non combined immunization group (Experimental): The non combined immunization group receive SARS-CoV-2 inactivated vaccine (Vero cell)(first dose) on day 0, Quadrivalent Influenza Vaccine on day 14 and SARS-CoV-2 inactivated vaccine (Vero cell)(second dose) on day 28.
  Interventions: Biological: Two doses of inactivated SARS-CoV-2 vaccine at the schedule of day 0,28 and one dose Quadrivalent Influenza Vaccine on day 14.

INTERVENTIONS:
Biological: Two doses of inactivated SARS-CoV-2 vaccine at the schedule of day 0,28 and one dose Quadrivalent Influenza Vaccine on day 0 or day 28. — The inactivated SARS-CoV-2 vaccine was manufactured by Sinovac Research & Development Co., Ltd., with a antigen content of 600SU/0.5ml. The Quadrivalent Influenza Vaccine manufactured by Sinovac Biotech Co.,Ltd. including 4 antigens H1N1, H3N2, BV and BY, 15μg for each, 0.5ml per dose.
  Arms: Combined immunization group
Biological: Two doses of inactivated SARS-CoV-2 vaccine at the schedule of day 0,28 and one dose Quadrivalent Influenza Vaccine on day 14. — The inactivated SARS-CoV-2 vaccine was manufactured by Sinovac Research & Development Co., Ltd., with a antigen content of 600SU/0.5ml. The Quadrivalent Influenza Vaccine manufactured by Sinovac Biotech Co.,Ltd. including 4 antigens H1N1, H3N2, BV and BY, 15μg for each, 0.5ml per dose.
  Arms: Non combined immunization group

SUMMARY:
This study is an open-label, single-center, randomized phase IV clinical trial of the SARS-CoV-2 inactivated vaccine manufactured by Sinovac Research & Development Co., Ltd. The purpose of this study is to evaluate the safety and immunogenicity of concomitant administration of the SARS-CoV-2 Inactivated Vaccine (Vero cell) with Quadrivalent Influenza Vaccine in adults aged from 18 to 59 Years

DETAILED DESCRIPTION:
This study is an open-label, single-center, randomized phase IV clinical trial of the SARS-CoV-2 inactivated vaccine (Vero cell) manufactured by Sinovac Research & Development Co., Ltd. The purpose of this study is to evaluate the safety and immunogenicity of concomitant administration of the SARS-CoV-2 Inactivated Vaccine (Vero cell) with Quadrivalent Influenza Vaccine in adults aged from 18 to 59 Years. 480 healthy adults as participants are randomly assigned into two groups in the ratio 1:1. The first group was the combined immunization group, which is randomly divided into two subgroups, 120 subjects in each group. The combined immunization subgroup Ⅰ receive SARS-CoV-2 inactivated vaccine &Quadrivalent Influenza Vaccine on day 0 and SARS-CoV-2 inactivated vaccine (second dose) on day 28.The combined immunization subgroup Ⅱ receive SARS-CoV-2 inactivated vaccine on day 0 and SARS-CoV-2 inactivated vaccine (second dose) & Quadrivalent Influenza Vaccine on day 28. The second group was the non combined immunization group，which receive SARS-CoV-2 inactivated vaccine (first dose) on day 0, Quadrivalent Influenza Vaccine on day 14 and SARS-CoV-2 inactivated vaccine (second dose) on day 28.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults aged 18-59 years;
* The subject can understand and voluntarily sign the informed consent form;
* Proven legal identity

Exclusion Criteria:

* Travel history / residence history of communities with case reports within 14 days;
* History of contact with a SARS-CoV-2 infection (positive in nucleic acid test) within 14 days;
* Have contacted patients with fever or respiratory symptoms from communities with case reports within 14 days;
* Two or more cases of fever and / or respiratory symptoms in a small contact area of volunteers, such as home, office etc. within 14 days;
* History of SARS-CoV-2 infection;
* History of asthma, history of allergy to the vaccine or vaccine components, or serious adverse reactions to the vaccine, such as urticaria, dyspnea, and angioedema;
* Congenital malformations or developmental disorders, genetic defects, severe malnutrition, etc.;
* Autoimmune disease or immunodeficiency / immunosuppression;
* Severe chronic diseases, severe cardiovascular diseases, hypertension and diabetes that cannot be controlled by drugs, liver or kidney diseases, malignant tumors, etc.;
* Severe neurological disease (epilepsy, convulsions or convulsions) or mental illness;
* Thyroid disease or history of thyroidectomy, spleenlessness, functional spleenlessness, spleenlessness or splenectomy resulting from any condition;
* Diagnosed abnormal blood coagulation function (eg, lack of blood coagulation factors, blood coagulopathy, abnormal platelets) or obvious bruising or blood coagulation;
* Immunosuppressive therapy, cytotoxic therapy, inhaled corticosteroids (excluding allergic rhinitis corticosteroid spray therapy, acute noncomplicated dermatitis superficial corticosteroid therapy) in the past 6 months;
* Physical examination has clinically significant abnormal hematology and biochemistry laboratory test results that exceed the reference value range (only applicable to phase I clinical trials):

  1. Blood routine test: white blood cell count, hemoglobin, platelet count;
  2. Detection of blood biochemical indicators: alanine aminotransferase (ALT), aspartate aminotransferase (AST), total bilirubin (TBIL), creatinine (CR), fasting blood glucose;
  3. Urine routine index: urine protein (PRO);
* History of alcohol or drug abuse;
* Receipt of blood products within in the past 3 months;
* Receipt of other investigational drugs in the past 30 days;
* Receipt of attenuated live vaccines in the past 14 days;
* Receipt of inactivated or subunit vaccines in the past 7 days;
* Acute diseases or acute exacerbation of chronic diseases in the past 7 days;
* Axillary temperature >37.0°C;
* Already pregnant (including a positive urine pregnancy test) or are breastfeeding, planning to get pregnant within 3 months;
* According to the investigator's judgment, the subject has any other factors that are not suitable for participating in the clinical trial.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 480 (Actual)
Dates: Start 2021-03-23 (Actual); Primary Completion 2021-05-28 (Actual); Study Completion 2021-05-28 (Actual)

PRIMARY OUTCOMES:
Safety index-incidence of adverse reactions within 7 days after each dose | Day 0-7 after each dose vaccination
  Incidence of adverse reactions within 7 days after each dose
Immunogenicity index-seroconversion rates of neutralizing antibody against SARS-CoV-2 | The 28th day after the second dose vaccination of the inactivated SARS-CoV-2 vaccine
  Neutralizing antibody assay will be performed using the micro-neutralization method. Seroconversion will be defined as a change from seronegative (<1:8) to seropositive (≥1:8), or ≥4 fold increase from baseline.

SECONDARY OUTCOMES:
Safety index-incidence of adverse reactions within 56 days after the first dose vaccination | Day 0-56 after the first dose vaccination
  Incidence of adverse reactions within 56 days after the first dose vaccination
Safety index-incidence of serious adverse events | Day 0-56 after the first dose vaccination
  SAE will be collected throughout the clinical trial.
Immunogenicity index-seropositive rates of neutralizing antibody against SARS-CoV-2 | The 28th day after each dose vaccination
  Neutralizing antibody assay will be performed using the micro-neutralization method, and subjects with a antibody titer ≥1:8 will defined as seropositive.
Immunogenicity index-geometric mean titer (GMT) of neutralizing antibody against SARS-CoV-2 | The 28th day after each dose vaccination
  Neutralizing antibody assay will be performed using the micro-neutralization method.
Immunogenicity index-geometric mean ratio (GMR) of neutralizing antibody against SARS-CoV-2 | The 28th day after each dose vaccination
  Neutralizing antibody assay will be performed using the micro-neutralization method. Ratio of post-vaccination titer divided by baseline titer will be calculated.
Immunogenicity index-seroconversion rates of influenza HI antibodies | The 28th day after the vaccination
  Seroconversion will be defined as a change from seronegative (<1:10) to protective (≥1:40), or ≥4 fold increase from baseline(≥1:10).
Immunogenicity index-protective rates of influenza HI antibodies | The 28th day after the vaccination
  The standard of reaching the protective rate is that the antibody titer ≥1:40.
Immunogenicity index-geometric mean titer (GMT) of influenza HI antibodies | The 28th day after the vaccination
  influenza HI antibodies assay will be performed using the micro hemagglutination inhibition test
Immunogenicity index-geometric mean ratio (GMR) of influenza HI antibodies | The 28th day after the vaccination
  influenza HI antibodies assay will be performed using the micro hemagglutination inhibition test

CONTACTS AND LOCATIONS:
Overall Officials: Huakun Lv, Master, Principal Investigator — Zhejiang Provincial Center for Disease Control and Prevention
Locations (1):
- Kaihua county Center for Disease Control and Prevention, Quzhou, Zhejiang, China